CLINICAL TRIAL: NCT02944656
Title: Gabapentin as an Adjunct to Paracervical Block for Perioperative Pain Management for Surgical Abortion: a Randomized Controlled Trial
Brief Title: Gabapentin as an Adjunct to Paracervical Block for Perioperative Pain Management
Acronym: Gaba
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Lisa Haddad, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00084198
Record Dates: First submitted 2016-10-13; First posted 2016-10-26 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Pain
Keywords: Perioperative pain; Outpatient surgery; Obstetrics/gynecology; Pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Gabapentin; gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gabapentin group (Experimental): This group will receive local anesthesia per clinic protocol plus Gabapentin 600mg 1-2 hours preoperatively.
  Interventions: Drug: Gabapentin
- Placebo group (Placebo Comparator): This group will receive local anesthesia per clinic protocol plus placebo 1-2 hours preoperatively.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Participants in this group will receive 600 mg of gabapentin given 1-2 hours pre-operatively in conjunction with perioperative paracervical block for surgical abortion. Gabapentin is an FDA approved medication that is used to prevent seizures and to treat various forms of chronic and acute pain.
  Other Names: Gaba; Neurontin
  Arms: Gabapentin group
Drug: Placebo — Participants in this group will receive 600 mg of gelatin capsules that are identical in appearance to gabapentin capsules. The placebo will be given 1-2 hours pre-operatively in conjunction with perioperative paracervical block for surgical abortion.
  Arms: Placebo group

SUMMARY:
This is a randomized controlled trial of gabapentin 600 mg compared to placebo given 1-2 hours preoperatively in conjunction with perioperative paracervical block for surgical abortion. The researchers hypothesize that adding gabapentin to local anesthesia will reduce perioperative and postoperative pain associated with surgical abortion. Additionally, the researchers hypothesize that gabapentin will reduce nausea, vomiting, anxiety, and consumption of pain medication.

DETAILED DESCRIPTION:
Project Summary

Justification for the project

One half of all pregnancies among American women are unintended, with nearly 4 in 10 ending in pregnancy termination by abortion. Elective abortions are among the most common outpatient surgical procedure, with an estimated 46 million performed worldwide annually. The management of pain is critical to patient care throughout the abortion experience since the vast majority of women will experience pain with the procedure. Patients are most affected by pain during paracervical block, cervical dilation, suction aspiration, and post operatively with uterine cramping. Innovation in pain control and reduction of anxiety, nausea and vomiting using a low cost, well-tolerated intervention could impact thousands of women each year.

Proposed research

This is a randomized controlled trial of gabapentin 600 mg compared to placebo given 1-2 hours preoperatively in conjunction with perioperative paracervical block for surgical abortion. The researchers hypothesize that adding gabapentin to local anesthesia will reduce perioperative and postoperative pain associated with surgical abortion. Additionally, the researchers hypothesize that gabapentin will reduce nausea, vomiting, anxiety, and consumption of pain medication.

New features

Gabapentin as an adjunct o pain management has proven beneficial in gynecological surgery. Its use in similar surgical settings as an adjunct to pain management regiments has proven to be beneficial. It is generally well tolerated, inexpensive, has minimal side effects, and few contraindications.

Problems anticipated

The high volume at the study clinic will benefit recruitment efforts, however, as the coordination of this study may potentially disrupt clinic flow there will be limits on daily recruitment. Postoperative follow-up may be challenging, thus to reduce the impact of loss to follow-up, most of the outcomes are measured on the same day as the procedure. Further, multiple contact approaches will be employed and a second incentive offered after completion of the postoperative assessment.

ELIGIBILITY:
Inclusion Criteria:

* Women >=18 years-old
* Presenting for a surgical abortion
* Fluency in English and able to provide informed consent
* Has a driver to take them home following the procedure

Exclusion Criteria:

* Allergy, sensitivity or contraindication to gabapentin
* Severe renal disease
* Currently using gabapentin or pregabalin
* Contraindication to outpatient abortion under local anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Haddad, MD, MS, MPH, Principal Investigator — Emory University
Locations (1):
- Atlanta Women's Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hailstorks TP, Cordes SMD, Cwiak CA, Gray BA, Ge L, Moore RH, Haddad LB. Gabapentin as an adjunct to paracervical block for perioperative pain management for first-trimester uterine aspiration: a randomized controlled trial. Am J Obstet Gynecol. 2020 Dec;223(6):884.e1-884.e10. doi: 10.1016/j.ajog.2020.06.011. Epub 2020 Jun 11. PMID 32534843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Atlanta Women's Center in Atlanta, Georgia. Enrollment began on December 8, 2016 and all study procedures concluded on June 26, 2018.
Pre-assignment Details: A total of 122 individuals were eligible and consented to participate in the study. Six withdrew prior to randomization and an additional 2 withdrew prior to beginning the study, resulting in 114 receiving the intervention.
Groups:
- Gabapentin Group: Participants receiving local anesthesia per clinic protocol plus two 300mg capsules of gabapentin 1-2 hours prior to the procedure.
- Placebo Group: Participants receiving local anesthesia per clinic protocol plus two 300mg capsules of a placebo to match gabapentin 1-2 hours prior to the procedure.
Period: Overall Study
Arm/Group | Gabapentin Group | Placebo Group
Started | 57 | 57
Completed Procedure Day | 54 | 57
Completed Day 1 Follow up | 47 | 47
Completed | 47 | 47
Not Completed | 10 | 10
Not completed — No longer eligible | 3 | 0
Not completed — Lost to Follow-up | 7 | 10

BASELINE CHARACTERISTICS:
Population: The baseline population includes participants completing all study procedures on the day of surgery.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin Group | Placebo Group | Total
Number analyzed (Participants) | 54 | 57 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (5.5) | 26.8 (5.5) | 26.01 (5.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 57 | 111
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 51 | 55 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Black/African American | 35 | 41 | 76
  White/Caucasian | 15 | 12 | 27
  Mixed or multi-racial | 0 | 4 | 4
  Other | 2 | 0 | 2
  Native Hawaiian/Pacific Islander | 0 | 0 | 0
  Don't know/Refused/Not Specified | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 54 | 57 | 111
Gestational age [Mean (Standard Deviation); unit: days] | 60.1 (15.1) | 62.5 (13.2) | 61.3 (14.10)

OUTCOME MEASURES:

1. Primary Outcome: Pain at Time of Uterine Evacuation
Description: The primary outcome measure is a pain score using a 100-mm visual analog scale (VAS) measured intraoperatively at time of evacuation. "No pain" is scored as 0 and "worst pain imaginable" is scored as 100.
Time Frame: During the procedure on Study Day 1
Population: Participants completing all assessments on the day of the procedure are included in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 54 | 57
score on a scale
  Paracervical block | 63.79 (3.77) | 62.21 (3.52)
  Dilation | 64.58 (3.74) | 66.12 (3.54)
  Aspiration | 67.77 (3.63) | 71.06 (3.49)

2. Secondary Outcome: Perioperative Pain Level
Description: Pain level at a variety of time points will be measured using a 100-mm visual analog scale (VAS) to log the change in pain levels between the study arms. "No pain" is scored as 0 and "worst pain imaginable" is scored as 100. Pain will be assessed immediately prior to the procedure, at completion of the procedure (removal of the speculum), 10 minutes following the procedure, and 30 minutes following the procedure (at discharge).
Time Frame: Pre-procedure through post-procedure on Study Day 1
Population: Participants completing all assessments on the day of the procedure are included in this analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 54 | 57
score on a scale
  Prior to procedure | 20.76 (3.60) | 22.48 (3.49)
  Speculum removal | 44.10 (3.60) | 47.61 (3.52)
  10 minutes post-procedure | 30.64 (3.65) | 43.68 (3.47)
  30 minutes post-procedure | 20.89 (3.68) | 31.65 (3.54)

3. Secondary Outcome: Number of Participants Using Pain Medication
Description: The number of participants reporting filling and using the prescription for ibuprofen postoperatively. During the follow-up phone call on the day after the procedure, participants were asked whether or not they filled the pain medication prescription and if they took any of the medication.
Time Frame: Postoperative Day 1
Population: Participants completing the follow up assessment one day after the procedure are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 47 | 47
Participants | 24 | 27

4. Secondary Outcome: Perioperative Nausea
Description: Nausea level was measured using a 100-mm visual analog scale (VAS) to log the change in nausea levels between the study arms. No nausea is reported as 0 while "worst nausea I have ever felt" is reported at 100. Nausea was reported immediately prior to the procedure, 10 minutes following the procedure, and 30 minutes following the procedure.
Time Frame: Pre-procedure through post-procedure on Study Day 1
Population: Participants completing all assessments on the day of the procedure are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 54 | 57
score on a scale
  Prior to procedure | 26 [3 to 57] | 26 [9 to 59]
  10 minutes post-procedure | 1 [0 to 22] | 12 [0 to 52]
  30 minutes post-procedure | 0 [0 to 16] | 5 [0 to 26]

5. Secondary Outcome: Perioperative Vomiting
Description: Participants reported if they vomited during the perioperative period to assess changes in vomiting incidences between the study arms. Vomiting is reported for the time periods of immediately prior to the procedure, 10 minutes following the procedure, and 30 minutes following the procedure.
Time Frame: Pre-procedure through post-procedure on Study Day 1
Population: Participants completing all assessments on the day of the procedure are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 54 | 57
Participants
  Prior to procedure | 4 | 7
  10 minutes post-procedure | 5 | 2
  30 minutes post-procedure | 5 | 5

6. Secondary Outcome: Anxiety Levels
Description: Participants reported how much anxiety they were currently experiencing on a 100-point scale where "No Anxiety" is scored as 0 and "Extremely Anxious" is scored as 100. Anxiety is reported for the time periods of immediately prior to the procedure, 10 minutes after the procedure, and 30 minutes after the procedure.
Time Frame: Pre-procedure through post-procedure on Study Day 1
Population: Participants completing all assessments on the day of the procedure are included in this analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 54 | 57
score on a scale
  Prior to procedure | 66 [21 to 83] | 72 [52 to 96.5]
  10 minutes post-procedure | 14 [0 to 36] | 17 [0 to 49]
  30 minutes post-procedure | 4 [0 to 29] | 2 [0 to 27]

7. Secondary Outcome: Side Effects
Description: Participants were asked if they experienced dizziness, lack of muscle control, sleepiness or drowsiness, weakness or lack of energy, headache, or visual changes.
Time Frame: 10 and 30 minutes post procedure on Study Day 1
Population: This analysis includes participants responding to the side effects questions. Two did not answer any questions. Two participants in the gabapentin group did not complete the side effect assessment at 30 minutes post-procedure. One participant in the placebo group did not respond to the assessment of weakness at 30 minutes post-procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 53 | 56
Participants
  Dizziness 10 minutes post-procedure | 27 | 23
  Dizziness 30 minutes post-procedure: number analyzed (Participants) | 51 | 56
  Dizziness 30 minutes post-procedure | 19 | 15
  Lack of muscle control 10 minutes post-procedure | 9 | 9
  Lack of muscle control 30 minutes post-procedure: number analyzed (Participants) | 51 | 56
  Lack of muscle control 30 minutes post-procedure | 5 | 10
  Sleepiness/drowsiness 10 minutes post-procedure | 38 | 34
  Sleepiness/drowsiness 30 minutes post-procedure: number analyzed (Participants) | 51 | 56
  Sleepiness/drowsiness 30 minutes post-procedure | 30 | 29
  Weakness 10 minutes post-procedure | 33 | 34
  Weakness 30 minutes post-procedure: number analyzed (Participants) | 51 | 55
  Weakness 30 minutes post-procedure | 20 | 28
  Headache 10 minutes post-procedure | 5 | 4
  Headache 30 minutes post-procedure: number analyzed (Participants) | 51 | 56
  Headache 30 minutes post-procedure | 4 | 4
  Vision changes 10 minutes post-procedure | 9 | 11
  Vision changes 30 minutes post-procedure: number analyzed (Participants) | 51 | 56
  Vision changes 30 minutes post-procedure | 3 | 5

8. Secondary Outcome: Moderate Pain at Postoperation Follow-up Assessment
Description: During the Postoperative Day 1 phone call, participants self reported how much they experienced moderate pain in the last 24 hours where 10 = none of the time and 0 = all of the time. "Moderate pain" was defined according to the perception of each participant.
Time Frame: Postoperative Day 1
Population: Participants completing the follow up assessment one day after the procedure are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 47 | 47
units on a scale | 5.2 (3.5) | 5.2 (3.4)

9. Secondary Outcome: Severe Pain at Postoperation Follow-up Assessment
Description: During the Postoperative Day 1 phone call, participants self reported how much they experienced severe pain in the last 24 hours where 10 = none of the time and 0 = all of the time. "Severe pain" was defined according to the perception of each participant.
Time Frame: Postoperative Day 1
Population: Participants completing the follow up assessment one day after the procedure are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 47 | 47
units on a scale | 3.5 (4.1) | 3.2 (4.1)

10. Secondary Outcome: Nausea or Vomiting at Postoperation Follow-up Assessment
Description: During the Postoperative Day 1 phone call, participants self reported how much they experienced nausea or vomiting in the last 24 hours where 10 = none of the time and 0 = all of the time. Nausea and vomiting were self-reported together as a single outcome.
Time Frame: Postoperative Day 1
Population: Participants completing the follow up assessment one day after the procedure are included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 47 | 47
units on a scale | 2.3 (3.9) | 3.2 (4.1)

11. Secondary Outcome: Vomiting Since Leaving Clinic
Description: During the Postoperative Day 1 phone call, participants self reported whether or not they had vomited since leaving the clinic.
Time Frame: Postoperative Day 1
Population: Participants completing the follow up assessment one day after the procedure are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 47 | 47
Participants
  No vomiting | 46 | 45
  Vomiting at least once | 1 | 2

12. Secondary Outcome: Overall Satisfaction With the Procedure
Description: Overall satisfaction with the procedure was assessed on a 10-point scale on the day after the procedure, where 1 = very dissatisfied and 10 = very satisfied.
Time Frame: Postoperative Day 1
Population: Participants completing the follow up assessment one day after the procedure are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin Group | Placebo Group
Number analyzed (Participants) | 47 | 47
Participants
  1 (very dissatisfied) | 0 | 1
  2 | 0 | 0
  3 | 0 | 2
  4 | 0 | 2
  5 | 5 | 4
  6 | 0 | 1
  7 | 4 | 2
  8 | 15 | 7
  9 | 5 | 11
  10 (very satisfied) | 18 | 17

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected from the time of investigational medication administration through the follow up phone call on the day after the procedure.
Description: In addition to specific side effects collected as an outcome measure, adverse effects were tracked and monitored during the study. An adverse event is defined as any health-related reaction, effect, toxicity or abnormal laboratory result experienced during the course of the study, irrespective of relationship to the study intervention.
Arm/Group | Gabapentin Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/57
Other Adverse Events (participants affected / at risk) | 1/54 | 1/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin Group (N=54) | Placebo Group (N=57)
Low Blood Pressure (General disorders) | 1 | 0
Increased nausea and vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT02944656/Prot_SAP_000.pdf